CLINICAL TRIAL: NCT03850795
Title: PROCADE: A Multinational Phase 3, Randomized, Double-Blind, Non-inferiority, Efficacy and Safety Study of Oral HC-1119 Versus Enzalutamide in Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: HC-1119 Versus Enzalutamide in Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated by Sponsor for various factors including prolonged duration and enrollment challenges
Sponsor: Hinova Pharmaceuticals USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC1119-CS-03
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer Metastatic; Castration-resistant Prostate Cancer
Keywords: HC-1119; enzalutamide
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HC-1119 (Experimental): Oral dose of 80 mg/day
  Interventions: Drug: HC-1119
- enzalutamide (Active Comparator): Oral dose of 160 mg/day
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: HC-1119 — oral once daily 80 mg
  Arms: HC-1119
Drug: Enzalutamide — oral once daily 160 mg
  Arms: enzalutamide

SUMMARY:
This study is a multinational Phase 3, randomized, double-blind, non-inferiority, efficacy and safety study of oral HC-1119 (80 mg/day) versus enzalutamide (160 mg/day) in asymptomatic or mildly symptomatic patients with progressive metastatic castration-resistant prostate cancer (mCRPC).

The following assessment of prostate cancer status will be collected during the course of the trial: soft tissue disease on computed tomography (CT) scan or on magnetic resonance imaging (MRI), bone disease on radionuclide bone scans, FACT-P and EQ-5D, Brief Fatigue Inventory, and PSA.

Throughout the study, safety and tolerability will be assessed by the recording of adverse events, monitoring of vital signs and physical examinations, safety laboratory evaluations, and 12-lead electrocardiograms (ECGs). Blood samples for population pharmacokinetics for HC-1119 and enzalutamide and related metabolites will be collected.

DETAILED DESCRIPTION:
This study is a multinational Phase 3, randomized, double-blind, non-inferiority, efficacy and safety study of oral HC-1119 (80 mg/day) versus enzalutamide (160 mg/day) in asymptomatic or mildly symptomatic patients with progressive metastatic castration-resistant prostate cancer (mCRPC). Patients must not have been previously treated with next generation AR-Inhibitors or Androgen-biosynthesis Inhibitors, or prior progression on ketoconazole.

The following assessments of prostate cancer status will be collected during the course of the trial: soft tissue disease on computed tomography (CT) scan or on magnetic resonance imaging (MRI), bone disease on radionuclide bone scans, FACT-P and EQ-5D, Brief Fatigue Inventory, and PSA. Radiographic disease progression is defined by the Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) for soft tissue disease, or the appearance of two or more new bone lesions on bone scan.

Throughout the study, safety and tolerability will be assessed by the recording of adverse events, monitoring of vital signs and physical examinations, safety laboratory evaluations, and 12-lead electrocardiograms (ECGs). Blood samples for population pharmacokinetics for HC-1119 and enzalutamide and related metabolites will be collected pre-dose on Day 1 and prior to dosing on Days 8 (Week 2), 15 (Week 3) and 22 (Week 4), 29 (Week 5), 57 (Week 9), 85 (Week 13) and Day 169 (Week 25). Blood samples for calculating a 24 hour pharmacokinetic profile of HC-1119 and enzalutamide and related metabolites will be collected in a subset of 24 Caucasian (non-Chinese) patients on Day 1 and at steady state in week 9.

Patients will have a safety follow-up visit 30 days after their last dose of study drug or prior to initiation of any new therapy, or an investigational agent, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following inclusion criteria:

1. Age 18 or older and willing and able to give informed consent.
2. Histologically or cytologically confirmed adenocarcinoma of the prostate without significant and relevant neuroendocrine differentiation or small cell features, per investigator's judgment.
3. Ongoing ADT with a GnRH analogue, antagonist or bilateral orchiectomy (i.e., surgical or medical castration).
4. For patients who have not had a bilateral orchiectomy, there must be a plan to maintain effective GnRH analogue or antagonist therapy for the duration of the trial.
5. Serum testosterone level < 1.7 nmol/L (50 ng/dL) at the Screening visit.
6. Patients receiving bisphosphonate or denosumab therapy must have been on stable doses for at least four weeks (from Day 1 visit).
7. Progressive disease at study entry defined as one or more of the following three criteria that occurred while the patient was on ADT as defined in eligibility criterion #3:

   1. PSA progression defined by a minimum of two rising PSA levels with an interval of ≥ 1 week between each determination. Patients who received an anti-androgen agent must have progression after withdrawal (≥ 4 weeks since last flutamide or ≥ 6 weeks since last bicalutamide or nilutamide). The PSA value at the Screening visit should be ≥ 2 µg/L (2 ng/mL)
   2. Soft tissue disease progression defined by RECIST 1.1
   3. Bone disease progression defined by PCWG3 with two or more new lesions on bone scan
8. Metastatic disease documented by measurable soft tissue disease by CT/MRI per RECIST 1.1 criteria. Patients are allowed to have any metastatic disease (i.e. bone metastasis) as long as they also have measurable soft tissue lesions per RECIST 1.1..
9. No prior cytotoxic chemotherapy for prostate cancer.
10. Asymptomatic or mildly symptomatic from prostate cancer.
11. ECOG performance status of 0-1 per the Investigators' clinical assessment
12. Estimated life expectancy of ≥ 6 months
13. Able to swallow the study drug and comply with study requirements
14. All sexually active patients are required to use a condom as well as meet 1 of the following:

    1. Patient is non-fertile (orchiectomy) or has a female partner of non-childbearing potential (i.e., post-menopausal, surgically sterilized, hysterectomy)
    2. Patient and his female partner must agree to use an adequate contraceptive method from the first day of dosing until 3 months after the last dose to prevent pregnancies. Adequate contraceptive method is defined as:

    i. Established use of oral, injected, or implanted hormonal methods of contraception.

    ii. Placement of an intra-uterine device or intra-uterine system. iii. Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.

    iv. Tubal ligation for at least 6 months prior to screening.
15. Male patient engaged in sexual activity with a pregnant female is required to use a condom from the first day of dosing until 3 months after the last dose of treatment with study drugs.

Exclusion Criteria:

Subjects must NOT meet any of the following exclusion criteria:

1. Severe concurrent disease, infection, or co-morbidity that, in the judgment of the investigator, would make the patient inappropriate for enrollment.
2. Known or suspected brain metastasis or active leptomeningeal disease.
3. Regular daily use of opiate analgesics for pain from prostate cancer within four weeks of enrollment (Day 1 visit).
4. WBC count < 3,000/µL, or absolute neutrophil count < 1,500/µL, or platelet count < 100,000/µL, or hemoglobin < 5.6 mmol/L (9 g/dL) at the Screening visit (NOTE: patients may not have received any growth factors or blood transfusions or any therapeutic invention within 14 days of the hematologic laboratory values obtained at the Screening visit).
5. Total bilirubin, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal at the Screening visit; no therapeutic invention within 14 days before screening.
6. Creatinine clearance < 30 mL/min as calculated using the Cockcroft-Gault equation at the Screening visit. Creatinine Clearance (mL/min) = [[140-Age (years)] * Weight (kg)] / [72 * Serum Creatinine (mg/dL)]
7. Albumin < 30 g/L (3.0 g/dL) at the Screening visit, no therapeutic invention within 14 days before screening.
8. History of another malignancy within the previous two years other than curatively treated non-melanomatous skin cancer.
9. Treatment with flutamide within four weeks of enrollment (Day 1 visit).
10. Treatment with bicalutamide or nilutamide within six weeks of enrollment (Day 1 visit).
11. Treatment with 5-α reductase inhibitors (finasteride, dutasteride), estrogens within four weeks of enrollment (Day 1 visit).
12. Treatment with systemic biologic therapy for prostate cancer (other than approved bone targeted agents) within four weeks of enrollment (Day 1 visit).
13. Use of herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (e.g., saw palmetto) or systemic corticosteroids greater than the equivalent of 10 mg of prednisone/prednisolone per day within four weeks of enrollment (Day 1 visit).
14. Prior use, or participation in a clinical trial, of an agent that blocks androgen synthesis (e.g., abiraterone) or blocks the AR (e.g., apalutamide, darolutamide, enzalutamide, proxalutamide).
15. Participation in a previous clinical trial of HC-1119.
16. Use of an investigational agent within four weeks of enrollment (Day 1 visit).
17. Radiation therapy for treatment of the primary tumor within three weeks of enrollment (Day 1 visit).
18. Radionuclide therapy (Radium 223) for treatment of metastasis within four weeks of enrollment (Day 1 visit).
19. Clinically significant cardiovascular disease or condition
20. Treatment with strong CYP2C8 inhibitors and inducers, CYP3A4 inducers, medications which are known to prolong the QT interval (see Appendix C).
21. History of seizure or any condition that may predispose to seizure.
22. Conditions that predispose subjects to increased risk for falls or fractures according to the discretion of the Investigator.
23. Gastrointestinal disorder affecting absorption (e.g., gastrectomy, active peptic ulcer disease within last three months).
24. Major surgery within four weeks prior to enrollment (Day 1 visit).
25. Have active infection with HBV measured by hepatitis B surface antigen (HBsAg) test, HCV measured by RNA test and HIV measured by antibody test.
26. Have known active tuberculosis.
27. Known hypersensitivity to HC-1119, enzalutamide, or any of the excipients.
28. Rare hereditary problems of fructose intolerance due to sorbitol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Week 24
  To determine the efficacy of HC-1119 as compared to enzalutamide as assessed by overall response rate (ORR) by RECIST 1.1.

SECONDARY OUTCOMES:
PSA decline of ≥50% from baseline | Week 24
  To determine the efficacy of HC-1119 as compared to enzalutamide as assessed by decline of ≥50% from baseline
Radiographic Progression-free Survival (rPFS) | Week 24
  To determine the efficacy of HC-1119 as compared to enzalutamide as assessed by radiographic progression-free survival (rPFS)
Overall Survival (OS) | Week 24
  To determine the efficacy of HC-1119 as compared to enzalutamide as assessed by overall survival (OS)
Safety and Tolerability (based on Common Terminology Criteria for Adverse Events (CTCAE), version 5.0) | Week 24
  To determine the safety and tolerability of orally administrated HC-1119 as compared to enzalutamide based on Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Locations (58):
- United States (8):
  - Urology Center of Colorado, 2777 Mile High Stadium Circle, Denver, Colorado
  - Urologic Surgeons of Washington, Washington D.C., District of Columbia
  - First Urology PSC, 101 Hospital Boulevard, Jeffersonville, Indiana
  - Clinical Research Solutions PC, Middleburg Heights, Ohio
  - MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Keystone Urology Specialists, Lancaster, Pennsylvania
  - Urology San Antonio Stone Oak, 18915 Meisner Drive, San Antonio, Texas
  - Providence Regional Cancer System, Lacey, Washington
- Australia (3):
  - Icon Cancer Care Gold Coast, Southport, Queensland
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Affinity Clinical Research, Nedlands
- Kepler Universitätsklinikum Linz, Linz, Austria
- Canada (2):
  - Fe/Male Health Centre, Oakville, Ontario
  - CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec
- Denmark (2):
  - Aalborg Universitetshospital, Aalborg
  - Odense Universitetshospital, Odense C
- Finland (4):
  - Helsinki University Hospital Comprehensive Cancer Center - PPDS, Helsinki
  - Oulun Yliopistollinen Sairaala, Oulu
  - Seinäjoen Keskussairaala, Seinäjoki
  - Tampereen yliopistollinen sairaala, Tampere
- France (6):
  - Hopital Foch, Suresnes, Hauts-de-Seine
  - Centre Jean Bernard Clinique Victor Hugo, Le Mans
  - CHRU Lille, Lille
  - Centre Léon Berard, Lyon
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hopital d'Instruction des Armées de Begin, Saint-Mandé
- Germany (4):
  - Urologische Studienpraxis, Nürtingen, Baden-Wurttemberg
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Tübingen, Tübingen
  - UroGynZentrum Wall, Wuppertal
- Italy (2):
  - Azienda Ospedaliera S Maria Di Terni, Terni, Umbria
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona
- Netherlands (4):
  - Canisius Wilhelmina Ziekenhuis, Nijmegen, Gelderland
  - Catharina Hospital, Eindhoven, North Brabant
  - Antonius Ziekenhuis, Sneek, Provincie Friesland
  - Hagaziekenhuis, The Hague, South Holland
- Poland (5):
  - Clinical Research Center Spolka z Ograniczona, Poznan, Greater Poland Voivodeship
  - NZOZ Centrum Urologiczne Sp zoo, Mysłowice, Silesian Voivodeship
  - Onko-Centrum Sp. z o.o., Lublin
  - Urologica Praktyka Lekarska Adam Marcheluk, Siedlce
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy, Warsaw
- Russia (7):
  - Altay Regional Oncology Center, Barnaul
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Federal State Institution Medical Radiology Research Center, Obninsk
  - Clinical Oncology Dispensary, Omsk
  - First St. Petersburg State Medical University n.a. I.P Pavlov, Saint Petersburg
  - GBUZ Saint Petersburg Clinical Research Center of Specialized Types of Care (Oncology), Saint Petersburg
  - Hospital Orkli LLC, Saint Petersburg
- Spain (6):
  - C.H. Regional Reina Sofia - PPDS, Córdoba
  - Hospital Lucus Augusti, Lugo
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Malaga - Hospital Civil, Málaga
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Fundacion Instituto Valenciano de Oncologia, Valencia
- United Kingdom (4):
  - Diana Princess of Wales Hospital, Grimsby, South Humberside
  - Belfast City Hospital, Belfast
  - Royal Marsden Hospital - London, London
  - Mount Vernon Hospital, Northwood

IPD SHARING:
Plan to Share IPD: No